CLINICAL TRIAL: NCT06519344
Title: An Exploratory Clinical Study Evaluating the Safety and Efficacy of Intravenous Anti-CD20/CD30-CAR-T Cell Infusion in Relapsed/Refractory Lymphoma Patients.
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Responsible Party: Principal Investigator, Aibin Liang，MD，Ph.D., professor,Chief Physician,Vice President of Tongji Hospital, Tongji University School of Medicine etc., Shanghai Tongji Hospital, Tongji University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD20/CD30-CN-A2
Record Dates: First submitted 2024-07-19; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: B Cell Malignancies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-CD20/CD30-CAR-T Cells (Experimental): anti-CD20/CD30-CAR-T cell infusion.Infusion doses:The planned infusion doses are follows：the first dose group at 3E5 cells/kg; the second dose group at 1E6 cells/kg; the third dose group at 3E6 cells/kg. Infusion doses refer to the number of CAR-positive cells.
  Administration method: anti-CD20/CD30-CAR-T cells are administered intravenously via an infusion pump at approximately 2-5 mL/minute, with a recommended infusion duration of less than 30 minutes.
  Interventions: Biological: anti-CD20/CD30-CAR-T Cells

INTERVENTIONS:
Biological: anti-CD20/CD30-CAR-T Cells — Before cell infusion,researchers may decide, based on necessity, whether to administer prophylactic medication,which may include options such as acetaminophen and diphenhydramine, or H1 antihistamines, among others. Subjects are allowed to receive adequate supportive care after anti-CD20/CD30-CAR-T cell infusion,including blood transfusions and blood products, antibiotic therapy, antiemetics, antidiarrheals, analgesice,etc.

SUMMARY:
This study is a single-center,open-label,single-dose clinical trial of anti-CD20/CD30-CAR-T cell therapy in relapsed/refractory B-cell tumor patients after lymphocyte depletion pre-treatment.

In this study phase,a traditional "3+3"trial design is employed for dose escalation.

DETAILED DESCRIPTION:
This study is a single-center, open-label, single-dose clinical trial of anti-CD20/CD30-CAR-T cell therapy in relapsed/refractory lymphoma patients after lymphocyte depletion pre-treatment.

The study aims to include patients with CD20/CD30 double-positive relapsed/refractory lymphomas, CD20-positive relapsed/refractory B-cell lymphomas (including patients who have relapsed after anti-CD19-CAR-T cell therapy), and CD30-positive Hodgkin lymphoma. Participants will undergo screening, peripheral blood mononuclear cell (PBMC) collection, and lymphocyte depletion pre-treatment before receiving a single infusion of anti-CD20/CD30-CAR-T cells.

Throughout the study, efficacy assessments will occur at baseline and at 4 weeks post-treatment, and subsequently at 3 months, 6 months, 9 months, and 12 months, until disease progression (PD), relapse, change of treatment regimen, death, intolerable toxicity, investigator decision, or voluntary withdrawal (whichever comes first).

Safety evaluations of anti-CD20/CD30-CAR-T cell therapy will be conducted according to the Common Terminology Criteria for Adverse Events (CTCAE, version 5.0) by laboratory tests, 12-lead electrocardiograms, vital signs, and physical examinations. Additionally, blood samples will be collected to assess cellular pharmacokinetics and explore the effects of cellular therapy on ferritin, C-reactive protein, and related cytokines.

The study is designed as an exploratory research project, subject to implementation conditions at the research center. Dose escalation during this study phase will follow a traditional "3+3" trial design.

ELIGIBILITY:
Inclusion Criteria:

(1) Voluntary participation in the clinical study; complete understanding by self or legally authorized guardian, informed of the study, and signing the Informed Consent Form (ICF); willing and able to comply with all trial procedures.

(2) Age between 18 and 70 years.

(3) Patients refractory or relapsed after current standard treatments (including allogeneic or autologous hematopoietic stem cell transplantation), and unsuitable for other treatment options such as second hematopoietic stem cell transplantation. Refractory/relapsed lymphoma is defined as:

1. No response to first-line therapy (primary refractory disease, excluding subjects intolerant to first-line therapy):

   - Progression of Disease (PD) assessment after first-line treatment
   * Best response of Stable Disease (SD) after at least 4 cycles of first-line treatment (e.g., 4 cycles of RCHOP), with SD maintenance duration not exceeding 6 months after the last dose.
2. No response to second-line or subsequent therapies:

   * PD as best response to the most recent treatment regimen
   * Best response of SD after at least 2 cycles of last-line treatment, with SD maintenance duration not exceeding 6 months after the last dose.
3. Refractory post autologous stem cell transplantation (ASCT):

   * Disease progression or relapse ≤12 months after ASCT (relapsing subjects must have biopsy-proven relapse)
   * If salvage therapy is performed post-ASCT, subjects must have had no response or relapse after the last-line treatment.
   * Relapsed or refractory disease after two or more lines of systemic therapy.

     (4) Lymphoma patients with target antigens meeting the following criteria:
   * CD20/CD30 double-positive lymphomas
   * Relapse after anti-CD19-CAR-T cell therapy, and CD20-positive lymphomas
   * Never received anti-CD19-CAR-T cell therapy, CD20-positive lymphomas
   * CD30-positive Hodgkin lymphoma.

     (5) Included lymphoma subtypes:
   * DLBCL-NOS (Diffuse Large B-Cell Lymphoma, not otherwise specified)
   * Primary mediastinal large B-cell lymphoma (PMBCL)
   * Transformed follicular lymphoma (TFL), previously treated with follicular lymphoma chemotherapy, subsequently transformed into DLBCL, refractory disease
   * Mantle cell lymphoma
   * High-grade B-cell lymphoma
   * Chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL)
   * Hodgkin lymphoma (HL).

     (6) ECOG performance status ≤2.

     (7) Expected survival of at least 12 weeks.

     (8) Adequate venous access (for single collection), and no other contraindications for blood cell separation.

     (9) Laboratory requirements at screening, with no hematologic evaluation within 7 days of receiving growth factors (long-acting granulocyte colony-stimulating factor (G-CSF/PEG-CSF) requires a 2-week interval):
   * Absolute neutrophil count ≥1.0×10^9/L;
   * Hemoglobin ≥60 g/L (without red blood cell transfusion within 7 days);
   * Platelets ≥50×10^9/L (CLL indication unrestricted);
   * Serum total bilirubin ≤1.5× upper limit of normal (ULN); or ≤3× ULN if liver tissue invasion by tumor;
   * Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤2.5× ULN, AST/ALT ≤5× ULN if liver tissue invasion by tumor;
   * Creatinine <1.5× ULN and estimated glomerular filtration rate ≥60 mL/minute.

     (10) Left ventricular ejection fraction ≥45%, echocardiogram (ECHO) showing no clinically significant pericardial effusion (excluding minimal or physiological effusions), and no clinically significant findings on electrocardiogram.

     (11) Baseline oxygen saturation >92% without supplemental oxygen.

     (12) Women of childbearing potential must have a negative serum or urine pregnancy test result (women who have undergone surgical sterilization or who are at least 2 years postmenopausal are not considered of childbearing potential).

Exclusion Criteria:

Here is the translation of the exclusion criteria for participants in a clinical study:

1. Evidence of central nervous system lymphoma on brain MRI; active primary central nervous system DLBCL, unless CNS involvement has been effectively treated (i.e., participant is asymptomatic) and there has been a local treatment interval of >4 weeks prior to enrollment.
2. Active central nervous system diseases such as epilepsy, cerebrovascular ischemia/hemorrhage, dementia, cerebellar diseases, or any autoimmune diseases with central nervous system involvement.
3. History of or concurrent malignancies other than CD19+ malignancies.
4. Clinically significant cardiac disease, or arrhythmias not controlled by medication.
5. Presence or suspicion of uncontrolled fungal, bacterial, viral, or other infections requiring intravenous antibiotics; simple urinary tract infections and uncomplicated bacterial pharyngitis are allowed.
6. Hepatitis B (positive hepatitis B surface antigen and hepatitis B DNA >1000 copies/mL) and hepatitis C (positive hepatitis C antibody).
7. Presence of any indwelling catheters or drainage tubes (e.g., percutaneous nephrostomy tube, Foley catheter, bile drainage tube, pleural/peritoneal/pericardial catheter); specialized central venous access devices like Port-A-Cath® or Hickman® catheters are allowed.
8. Use of the following medications prior to:

1) Ibrutinib within 1 day before apheresis. 2) Idelalisib (oral PI3Kδ inhibitor) within 2 days before apheresis. 3) Short-acting targeted therapy (such as tyrosine kinase inhibitors) within 72 hours before apheresis.

4) Venetoclax (BCL-2 inhibitor) within 4 days before apheresis. 5) Long-acting growth factors (such as pegfilgrastim) within 14 days before apheresis, or short-acting growth factors or mobilizing agents (such as granulocyte colony-stimulating factor (G-CSF)/filgrastim) within 5 days before apheresis.

6) Pharmacologic doses of corticosteroid therapy (>5 mg/day prednisone or equivalent) and other immunosuppressive drugs within 7 days before enrollment.

7) Radiotherapy within 14 days before enrollment. 8) Systemic cytotoxic drugs within 14 days before enrollment, including daily or weekly low-dose maintenance chemotherapy (e.g., cyclophosphamide, fludarabine, bendamustine, chlorambucil, methotrexate, vinblastine).

If bridging therapy is administered post-apheresis, there must be at least a 7-day interval between bridging therapy and CAR-T cell infusion.

9) Anti-PD1 or anti-PDL1 therapy within 4 weeks before enrollment. 10) Vaccination within 4 weeks before enrollment. 11) Donor lymphocyte infusion (DLI) within 4 weeks before enrollment. 12) Immunostimulatory or immunosuppressive therapy within 3 months before enrollment (such as interferon-α, interferon-β, IL-2, lenalidomide, efalizumab, alemtuzumab, cyclosporine, or methotrexate).

(9) Active graft-versus-host disease (GVHD) using the CIBMTR acute GVHD grading system ≥ grade 2 or requiring systemic steroids greater than physiological doses.

(10) History in the past 2 years of autoimmune diseases causing end-organ damage or requiring systemic immunosuppressive/disease-modifying agents, such as Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus.

(11) History in the past 12 months of myocardial infarction, cardiac vascular procedures or stent implantation, unstable angina, or other clinically significant cardiac diseases.

(12) History of genetic syndromes with bone marrow failure, such as Fanconi anemia, Costello syndrome, Shwachman-Diamond syndrome.

(13) Symptomatic deep vein thrombosis or pulmonary embolism requiring systemic anticoagulation therapy within 6 months before enrollment. Subjects requiring prophylactic anticoagulation are allowed.

(14) History of concurrent or prior malignancies (excluding basal cell carcinoma of the skin, in situ carcinoma of the breast/cervix, and other malignancies effectively controlled without treatment within the past five years).

(15) Use of other investigational medicinal products within 30 days before screening.

(16) Pregnant or lactating women of childbearing potential. Women who have undergone surgical sterilization or who are at least 2 years postmenopausal are not considered of childbearing potential.

(17) Participants unwilling to use contraception from agreeing to treatment until completion of lymphocyte depletion chemotherapy or CAR-T cell infusion within 12 months (whichever is longer).

(18) Any medical activities that could potentially interfere with the safety or efficacy evaluation of the study treatment.

(19) According to the investigator's judgment, participants who are unlikely to complete all study visits or procedures required by the protocol (including follow-ups), or comply with the requirements of participating in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-07-31 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity | Up to 28 days from CAR-T infusion
  The proportion of patients receiving CAR-T cells who encounter dose-limiting toxicities(DLTs). Safety evlauations are performed in accordance with the NCI-CTCAE version 5.0 standards(Cytokine Release Syndrome and neurotoxicity will be graded based on ASTCT/ASBMT grading criteria).

CONTACTS AND LOCATIONS:
Overall Officials: Aibin Liang, Principal Investigator — Shanghai Tongji Hospital, Tongji University School of Medicine

IPD SHARING:
Plan to Share IPD: No